CLINICAL TRIAL: NCT00061360
Title: A Randomized Trial of a Novel Immunosuppressive Combination of ATG, CsA and Sirolimus (Rapamune) vs a Slow Taper Cyclosporine Regimen in Subjects With Severe Aplastic Anemia
Brief Title: Improving Immunosuppressive Treatment for Patients With Severe Aplastic Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 030193; 03-H-0193
Record Dates: First submitted 2003-05-23; First posted 2003-05-26 (Estimated); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Severe Aplastic Anemia
Keywords: Bone Marrow Failure; Cyclosporine; Anti Thymocyte Globulin; Severe Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic; Bone Marrow Failure Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATG+CsA (Experimental): ATG+CsA for 6 months followed by a slow CsA taper in the subsequent 18 months
  Interventions: Drug: ATG+cyclosporine
- ATG+CsA+RA (Experimental): ATG+CsA+RAPA for 6 months
  Interventions: Drug: ATG+Rapamune+cyclosporine

INTERVENTIONS:
Drug: ATG+Rapamune+cyclosporine — ATG+Rapamune+cyclosporine
  Arms: ATG+CsA+RA
Drug: ATG+cyclosporine — ATG+cyclosporine
  Arms: ATG+CsA

SUMMARY:
Severe aplastic anemia (SAA) is a life-threatening bone marrow failure disorder characterized by pancytopenia and a hypocellular bone marrow. Allogeneic bone marrow transplantation and immunosuppressive treatment with anti-thymocyte globulin (ATG) and cyclosporine (CsA) have dramatically changed the natural course of this illness, with 5 year survival of 75% in patients undergoing either treatment. Since most patients are not suitable candidates for hematopoietic stem cell transplantation (HSCT) due to advanced age or lack of a histocompatible sibling, efforts at NHLBI have focused on improving immunosuppression treatment in order to improve response rates, survival, and to decrease relapse.

In our experience of 122 patients treated at NHLBI with the combination of ATG and cyclosporine, one quarter to one third did not respond; about 50% of responders relapsed; and 5 year survival was correlated with the robustness in blood cell count improvement at 3 months (reticulocyte or platelet count greater than or equal to 50,000 /uL). Why some patients do not respond initially while others relapse is unclear. Autoreactive T cells may be resistant to the effect of ATG/CsA (nonresponders), while in others residual autoreactive T cells expand post-treatment leading to hematopoietic stem cell destruction and recurrent pancytopenia (relapse). Therefore, novel immunosuppressive regimens to increase response rates and hematologic recovery at 3 months and to decrease relapse rates are needed. An ongoing NHLBI trial, which is close to completing accrual, has added mycophenolate mofetil (MMF) for a total of 18 months to standard ATG + CsA in an attempt to reduce the relapse rate after cyclosporine is discontinued. Preliminary results have been disappointing, with no marked reduction in relapse among patients who received MMF.

Sirolimus (rapamycin, Rapamune , RAPA) is a novel immunosuppressive agent, which acts synergistically with cyclosporine by blocking T cell activation through CsA-resistant pathways. The potentiation of the combination of CsA-RAPA has been established in vitro and in the clinical setting, mainly in islet cell and solid organ transplantation. The significant increase in response rate seen with the addition of CsA to ATG indicated that an inhibitory effect on T lymphocytes is important in blocking autoreactive T cells in aplastic anemia. The combination of CsA-RAPA may further block activated autoreactive T cells and therefore lead to improved response rates (and survival) and decreased relapse rates.

This prospective randomized phase II study will investigate two different immunosuppressive regimens in patients with severe aplastic anemia who have not received prior immunosuppressive therapy. One arm will receive ATG + CsA in addition to sirolimus for 6 months, and the second arm will receive standard ATG + CsA for 6 months followed by a slow taper of CsA with a 25% dose reduction every 3 months for the subsequent 18 months. This trial will determine the effectiveness of sirolimus in patients with aplastic anemia as well as the role of a cyclosporine taper in preventing relapses. Primary endpoint will be no longer meeting criteria for severe aplastic anemia while secondary endpoints are relapse, robustness of hematologic recovery at 3 months, survival, clonal evolution to PNH, myelodysplasia and acute leukemia.

10/11/2005. The Sirolimus (Rapamune) arm of the trial was stopped for lack of efficacy. The study will continue as a single arm study to establish if slow taper of CsA prevents relapse rates after initial standard treatment with ATG followed by CsA for six months.

DETAILED DESCRIPTION:
Severe aplastic anemia (SAA) is a life-threatening bone marrow failure disorder characterized by pancytopenia and a hypocellular bone marrow. Allogeneic bone marrow transplantation and immunosuppressive treatment with anti-thymocyte globulin (ATG) and cyclosporine (CsA) have dramatically changed the natural course of this illness, with 5 year survival of 75% in patients undergoing either treatment. Since most patients are not suitable candidates for hematopoietic stem cell transplantation (HSCT) due to advanced age or lack of a histocompatible sibling, efforts at NHLBI have focused on improving immunosuppression treatment in order to improve response rates, survival, and to decrease relapse.

In our experience of 122 patients treated at NHLBI with the combination of ATG and cyclosporine, one quarter to one third did not respond; about 50% of responders relapsed; and 5 year survival was correlated with the robustness in blood cell count improvement at 3 months (reticulocyte or platelet count greater than or equal to 50,000 /uL). Why some patients do not respond initially while others relapse is unclear. Autoreactive T cells may be resistant to the effect of ATG/CsA (nonresponders), while in others residual autoreactive T cells expand post-treatment leading to hematopoietic stem cell destruction and recurrent pancytopenia (relapse). Therefore, novel immunosuppressive regimens to increase response rates and hematologic recovery at 3 months and to decrease relapse rates are needed. An ongoing NHLBI trial, which is close to completing accrual, has added mycophenolate mofetil (MMF) for a total of 18 months to standard ATG + CsA in an attempt to reduce the relapse rate after cyclosporine is discontinued. Preliminary results have been disappointing, with no marked reduction in relapse among patients who received MMF.

Sirolimus (rapamycin, Rapamune , RAPA) is a novel immunosuppressive agent, which acts synergistically with cyclosporine by blocking T cell activation through CsA-resistant pathways. The potentiation of the combination of CsA-RAPA has been established in vitro and in the clinical setting, mainly in islet cell and solid organ transplantation. The significant increase in response rate seen with the addition of CsA to ATG indicated that an inhibitory effect on T lymphocytes is important in blocking autoreactive T cells in aplastic anemia. The combination of CsA-RAPA may further block activated autoreactive T cells and therefore lead to improved response rates (and survival) and decreased relapse rates.

This prospective randomized phase II study will investigate two different immunosuppressive regimens in patients with severe aplastic anemia who have not received prior immunosuppressive therapy. One arm will receive ATG + CsA in addition to sirolimus for 6 months, and the second arm will receive standard ATG + CsA for 6 months followed by a slow taper of CsA with a 25% dose reduction every 3 months for the subsequent 18 months. This trial will determine the effectiveness of sirolimus in patients with aplastic anemia as well as the role of a cyclosporine taper in preventing relapses. Primary endpoint will be no longer meeting criteria for severe aplastic anemia while secondary endpoints are relapse, robustness of hematologic recovery at 3 months, survival, clonal evolution to PNH, myelodysplasia and acute leukemia.

10/11/2005. The Sirolimus (Rapamune) arm of the trial was stopped for lack of efficacy. The study will continue as a single arm study to establish if slow taper of CsA prevents relapse rates after initial standard treatment with ATG followed by CsA for six months.

3/2/2006. The protocol was closed to new accrual.

ELIGIBILITY:
* INCLUSION CRITERIA:

Severe aplastic anemia confirmed at NIH by:

1. . Bone marrow cellularity less than 30% (excluding lymphocytes)
2. . At least two of the following: Absolute neutrophil count less than 500/ uL; Platelet count less than 20,000/ uL; Absolute reticulocyte count less than 60,000/ uL

Age greater than or equal to 2 years old

Weight greater than 12 kg

EXCLUSION CRITERIA:

Serum creatinine greater than 2.5 mg/dL

Underlying carcinoma (except local cervical, basal cell, squamous cell)

Prior immunosuppressive therapy with ATG, ALG, or high dose cyclophospamide.

Current pregnancy or lactation or unwillingness to take oral contraceptives or use an effective method of birth control.

Diagnosis of Fanconi anemia or other congenital bone marrow failure syndromes

Evidence of a clonal disorder on cytogenetics. Patients with super severe neutropenia (ANC less than 200/uL) will not be excluded if results of cytogenetics are not available or pending.

Underlying immunodeficiency state including seropositivity for HIV

Inability to understand the investigational nature of the study or give informed consent

Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient s ability to tolerate protocol therapy, or that death within 7-10 days is likely.

Ages: 2 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2003-06-26 (Actual); Primary Completion 2006-02-15 (Actual); Study Completion 2015-09-08 (Actual)

PRIMARY OUTCOMES:
Hematologic recovery in patients with severe aplastic anemia treated with a novel immunosuppressive combination of ATG, CsA and sirolimus. | 2 yrs
  Up to 10/11/2005- Response rate at 3 months defined as no longer meeting criteria for SAAFrom 10/11/2005-relapse rates after initial standard treatment with ATG followed by CsA for six months

SECONDARY OUTCOMES:
6-month response rate | 6 months
Robustness of hematologic recovery with reticulocyte count or platelet count 50,000/uL at 3 months | 3 months
Relapse | Ongoing
Clonal evolution to MDS, PNH or acute leukemia | Ongoing
Survival | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Neal S Young, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Zaimoku Y, Patel BA, Adams SD, Shalhoub R, Groarke EM, Lee AAC, Kajigaya S, Feng X, Rios OJ, Eager H, Alemu L, Quinones Raffo D, Wu CO, Flegel WA, Young NS. HLA associations, somatic loss of HLA expression, and clinical outcomes in immune aplastic anemia. Blood. 2021 Dec 30;138(26):2799-2809. doi: 10.1182/blood.2021012895. PMID 34724566
- [Derived] Scheinberg P, Wu CO, Nunez O, Scheinberg P, Boss C, Sloand EM, Young NS. Treatment of severe aplastic anemia with a combination of horse antithymocyte globulin and cyclosporine, with or without sirolimus: a prospective randomized study. Haematologica. 2009 Mar;94(3):348-54. doi: 10.3324/haematol.13829. Epub 2009 Jan 30. PMID 19181786
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2003-H-0193.html